CLINICAL TRIAL: NCT05579418
Title: The Safety and Long-Term Clinical Benefit of PCSK9i in Addition to Statin Therapy in Patients With ST-Segment Elevation Myocardial Infarction. A Randomized, Open Label Study.
Brief Title: The Safety and Long-Term Clinical Benefit of PCSK9i in STEMI Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Mohammed Thamer Ali, Consultant Interventional Cardiologist, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-22-366
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: STEMI; Dyslipidemias
Keywords: STEMI; PCSK9i; Evolocumab; Statin
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Dyslipidemias | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: The study is an investigator-initiated, prospective, randomized, open-label study. All patients presenting with STEMI will be screened for the trial, those patients with LDL-C levels higher than guideline-recommended targets despite prior high-intensity statin therapy, or when the LDL-C not projected to decrease below the recommended targets if they are newly initiated on high intensity statin therapy, will be considered for the study.
  Participants will be randomly assigned using permuted block design with a computer random number generator, the block size is fixed (8 per block) with random allocation within the block to either the control group or the interventional group (4 for each group, patient allocation within the block is randomly assigned). Once the patient has given consent to be included in the trial, he/she is then irreversibly randomized by opening the next sealed envelope, within the current block, containing his/her assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Active Comparator): Patient that qualify for the trial will be randomized for receiving the PCSK9i injection in addition to the standard medical therapy.
  Interventions: Drug: Evolocumab
- Control Arm (No Intervention): Patient will only receive the standard medical therapy, No PCSK9i

INTERVENTIONS:
Drug: Evolocumab — Evolocumab is an injection for management of dyslipidemia
  Other Names: Repatha
  Arms: Interventional Arm

SUMMARY:
Patients with acute coronary syndromes (ACS) have an increased risk of recurrent ischemic events, particularly during the first year following the index event, which is mainly due to unattended risk factors and/ or poor compliance with medications. Lowering low-density lipoprotein cholesterol (LDL-C) reduces cardiovascular morbidity and mortality in patients with atherosclerotic cardiovascular disease (ASCVD), with a magnitude of clinical benefit that is proportional to the reduction in LDL-C levels. Proprotein convertase subtilisin/ kexin type 9 (PCSK9) antibodies have emerged as a new class of drugs that rapidly and effectively lower LDL-C levels up to 77 % of the original value in combination with statins.

The primary objective of this study is to confirm the safety and the long-term clinical benefit associated with the use of PCSK9i when combined with statin in patients with ACS-STEMI.

The study is an investigator-initiated, prospective, randomized, open label study that will be the first study looking for the safety and the clinical benefit and outcome associated with the use of PCSK9i in ACS-STEMI patients specifically. Internationally, this will be the first trial studying the effect of PCSK9i on patients with acute myocardial infarction (STEMI) in terms of reduction in cholesterol level and reduction in cardiac events rate (re-infarction and cardiac death) after myocardial infarction. This trial will have a significant impact in the management of patients with STEMI, locally and internationally and it will be conducted purely in Qatar. This trial will help to improve the clinical outcome of patients in Qatar in terms of reduction of myocardial reinfarction rate and mortality.

DETAILED DESCRIPTION:
The study is an investigator-initiated, prospective, randomized, open-label study. Patients will be eligible for participation in the trial if they are between 18-70 years of age. All patients presenting with STEMI will be screened for the trial, those patients with LDL-C levels higher than guideline-recommended targets despite prior high-intensity statin therapy (on statin therapy prior to hospital admission), or when the LDL-C not projected to decrease below the recommended targets if they are newly initiated on high intensity statin therapy, will be considered for the study.

Procedures and study interventions.

1. Patients hospitalized for ST-segment elevation myocardial infarction [STEMI] with symptom onset <12 h prior to hospitalization) will be potentially eligible.
2. Patient will receive the standard care as per the HH guidelines in terms of coronary angiogram, standard therapy of statin, dual antiplatelet, B -Blockers and ACE.
3. These patients will be screened for suitability to participate in the study
4. The patients will be considered for enrolment if he/she is hemodynamically stable and had a successful PPCI to De-novo lesion in an infarct related artery (NOT stent thrombosis- those will be excluded from the study, also acute occlusion of cardiac grafts will be excluded from the study as well).
5. LDL- C will be assessed immediately post angiography: The patient will be eligible for the trial if the LDL-C levels at the screening blood test is one of the following:

   >1.8 mmol/l if patients are on stable (unchanged for >4 weeks before screening) treatment with high-intensity statin.

   2.3 mmol/l in patients previously taking low- or moderate-intensity statin. 3.2 mmol/l in patients not on statin treatment.
6. Eligible patients will be randomly assigned in a 1:1 ratio to one of the two groups: The control group or the intervention group.
7. The control group will receive the standard, guidelines directed optimal medical therapy.
8. The interventional group will receive Evolocumab 140 mg every 2 weeks in addition to the standard, guideline directed, optimal medical therapy.
9. The optimal medical therapy will include high intensity statin (either atorvastatin 40-80 mg/day or rosuvastatin 20-40 mg /day throughout the study) or maximal tolerated statin (in both groups the statin dose can be titrated up or down as per the standard clinical practice).
10. The study drug will be administered at baseline as early as possible but within 24 hr following hospitalization. In our institute, patients admitted with STEMI will receive primary percutaneous intervention by default. The average time for door to balloon time is around 50 minutes (department data). Randomization and drug administration is not possible within such a short time, in addition consider randomization and drug administration before angiography may results in delay of delivering standard therapy which is of not in the best interest of the patient.
11. The randomization will be done immediately after angiography and aim for drug administration within 24 hr of admission.
12. Blood samples will be obtained at baseline for assessment of fasting lipids and inflammatory markers.
13. All patients recruited for the trial, will receive medical treatment for ACS as per the Heart hospital and international guidelines. Patients that will be considered for the trial should have received coronary angiography and revascularization (percutaneous coronary intervention) as per the hospital guidelines.
14. Patients not fit or rejected re-vascularization with PCI or patient that will need coronary artery bypass grafting [CABG] surgery) will be excluded from this study.
15. Written informed consent will be obtained from all the patients.
16. The research team may ask for supervised injection when suspect non-compliance.

Information and investigation that will be collected from patient:

1. Patient will have blood test: Lipid panel, Liver function, and CRP will be done at 0,1, 2, 6 and 12, 18, and 24 months.
2. Carotid intimal thickening measurement: at 0, 6, 12, 24 months
3. Echocardiogram: 1,6,12,24 months
4. OPD Review for clinical evaluation: medication side effect, Chest pain, hospitalization or unplanned PCI at 1,2,3,6,12,18,24 months.

Randomization:

Participants will be randomly assigned using permuted block design with a computer random number generator, the block size is fixed (8 per block) with random allocation within the block to either the control group or the interventional group. of the patients (4 for each group, patient allocation within the block is randomly assigned). Once the patient has given consent to be included in the trial, he/she is then irreversibly randomized by opening the next sealed envelope, within the current block, containing his/her assignment.

The production of computer-generated sets of random allocations will be done by a research support unit (who will not be performing data collection) in advance of the start of the study.

Sample size calculation:

Our study is designed as a superiority trial powered for the primary endpoint. The average LDL-D cholesterol of patients admitted with ACS-STEMI to the Heart Hospital was 3.4 mmol based on calculating the average LDL-C of 150 patients with ACS-STEMI in the past 6 months (department Data).

Bases on the EVOPACS study above, statin alone therapy will reduce the LDL-C by 35 % (1.19 mmol), while Evolocumab + statin combination therapy will reduce LDL-C by 77 % (2.61 mmol). Expectations for cholesterol-lowering trials were set by the Cholesterol Treatment Trialists' Collaborators, who reported in 2005 that for each 1 mmol/L (38.6 mg/dL) reduction in LDL-C, cardiovascular events were reduced by a mean of 22%. Based on this, the expected reduction in cardiovascular event is 26 % with statin therapy alone and 57 % with Evolocumab + statin. Assuming 1000 cases of ACS-STEMI present to our emergency department every year, and event rate of 17-33 % post STEMI patient for those on moderate to high intensity statins at one year, 90 % power and 5 % significance level, the sample size was 144 for each arm. Accounting for the nature of the country of high travel and dropout nature, 20 % drop rate was added to the sample size, the final sample size for this trial was up rounded to 350 patients (originally was 346).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion and exclusion criteria:

Inclusion Criteria

* Male or female ≥ 18 years of age and less than 80 years
* Hospitalized for a recent ACS-STEMI within 12 hours of onset of symptoms.
* Successful revascularization with PCI.
* LDL-C levels defined as follows:

  * LDL-C ≥1.8 mmol/L in patients who have been receiving stable treatment with high-intensity statin within ≥ 4 weeks prior to enrollment (i.e., continuous treatment that has not changed with regard to statin intensity over the past 4 weeks)
  * LDL-C ≥2.3 mmol/L in patients who have been receiving stable treatment with low- or moderate-intensity statin within ≥ 4 weeks prior to enrollment (i.e., continuous treatment that has not changed with regard to statin intensity over the past 4 weeks)
  * LDL-C ≥3.2 mmol/L in patients who are statin-naïve or have not been on a stable (unchanged) statin regimen for at least 4 weeks prior to enrollment.
* Ability to understand the requirements of the study and to provide informed consent

Exclusion criteria

* Unstable clinical status (hemodynamic or electrical instability)
* Uncontrolled cardiac arrhythmia, defined as recurrent and symptomatic ventricular tachycardia or atrial fibrillation or flutter with rapid ventricular response not controlled by medications in the past 3 months prior to screening
* Severe renal dysfunction, defined by estimated glomerular filtration rate <30 ml/min/1.73m2
* Active liver disease or hepatic dysfunction, either reported in patient medical record or defined by aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels > 3x the upper limit of normal.
* Patient need urgent CABG
* patients symptoms onset is more than 12 hours.
* Reported intolerance to atorvastatin (any dose) OR statin intolerance defined by the following criteria:

  * inability to tolerate at least 2 different statins (one statin at the lowest starting average daily dose and the other statin at any dose).
  * intolerance associated with confirmed, intolerable statin-related adverse effect(s) or significant biomarker abnormalities.
  * symptom or biomarker changes resolution or significant improvement upon dose decrease or discontinuation.
* Known allergy to contrast medium, heparin, aspirin, ticagrelor or prasugrel
* Known sensitivity to any substances or medication to be administered during the trial
* Patients who previously received Evolocumab or other PCSK9 inhibitor
* Treatment with systemic steroids or systemic cyclosporine in the past 3 months.
* Known active infection or major hematologic, metabolic, or endocrine dysfunction in the judgment of the Investigator
* Patients who will not be available for study-required procedures in the judgment of the Investigator
* Current enrollment in another investigational device or drug study
* Active malignancy requiring treatment
* Pregnant women. For female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy, pregnancy is excluded by a pregnancy test prior to inclusion in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular events, defined as the composite of cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization. | 12 months
  The primary objective of this study is to confirm the safety and the long-term clinical benefit associated with the use of PCSK9i in combination with statin in patients with ACS-STEMI. The long terms clinical benefit is the reduction in major cardiovascular events, defined as the composite of cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization.
The safety of PCSK9i in patients with STEMI | 12 months
  The safety of PCSK9i use in patients admitted with STEMI in terms of adverse events and complications related to the use of PCSK9i.

SECONDARY OUTCOMES:
Percentage change in calculated LDL-C from baseline to end of study period. | 12 months
  The changes noted in the LDL-C levels from baseline ( time of recruitment) to end of study period.
Changes in carotid intimal thickening from baseline to the end of study period | 12 months
  The intima-medial thickness of common carotid artery will evaluated by B-mode ultrasound imaging, the delta changes in the carotid intima-medial thickness will be calculated.
Adverse events and serious adverse events reported during study period. | 12 months
  Any adverse events whether expected or not expected will be record and tabulated. These adverse events will be compared with the control group.
Changes in High-sensitivity C-reactive protein from baseline to the end of study period | 12 months
  Changes in High-sensitivity C-reactive protein from baseline to the end of study period
Changes in left ventricular ejection fraction from baseline to the end of study period . | 12 months
  Changes in left ventricular ejection fraction from baseline to the end of study period will be measured using echocardiogram.
Individual major cardiovascular events, defined as the composite of cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization. | 12 months
  The effect of PCSK9i use in STEMI patients for each of the outcome individually including: cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Ali, MD, Principal Investigator — Hamad Medical Corporation

IPD SHARING:
Plan to Share IPD: Yes
All patients details will be stored in an electronic database and will be shared if a request submitted to institution research board and approved.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 10 years
Access Criteria: Request has to be approved by PI and Heart Hospital Research Advisory Board.